CLINICAL TRIAL: NCT03757455
Title: Enhanced Recovery Versus Standard Recovery After Low-risk Pancreatoduodenectomy Identified With Acinar Cell Count or Total Pancreatectomy: a Randomized Controlled Trial
Brief Title: ERAS Protocol in Pancreaticoduodenectomy and Total Pancreatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enought participants
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18125
Record Dates: First submitted 2018-11-13; First posted 2018-11-29 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Cancer; Surgery--Complications; Pancreatic Fistula; Delayed Gastric Emptying; Pancreatic Hemorrhage
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula; Gastroparesis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enchanced recovery after surgery protocol (Experimental): ERAS-protocol as described in low risk patients after pancreaticoduodenectomy or total pancreatectomy
  Interventions: Procedure: ERAS protocol preoperative actions; Procedure: ERAS protocol intraoperative actions; Procedure: ERAS protocol postoperative actions
- Standard protocol (No Intervention): Standard recovery protocol after pancreaticoduodenectomy or total pancreatectomy

INTERVENTIONS:
Procedure: ERAS protocol preoperative actions — First appointment:
  - Enlightenment on the benefits and objectives of the ERAS protocol
  Call to the patient day before the surgery:
  Discussing the course, benefits and goals of care in ERAS 4 dl PreOp drink before bedtime
  Operation day:
  Fluid intake allowed 2 hours before surgery 2 dl PreOP drink 2 h before cutting
  Arms: Enchanced recovery after surgery protocol
Procedure: ERAS protocol intraoperative actions — Intraoperative:
  Drains in the peripancreatic or perihepatic regions are not set unless the surgeon sees this particular reason The nasogastric tube is removed at the end of the surgery
  Arms: Enchanced recovery after surgery protocol
Procedure: ERAS protocol postoperative actions — Postoperatively:
  Mobilization with nurses assisted Drinks allowed after 4h surgery
  POP 1:
  Drinking and normal food Removal of urinary catheter Intravenous liquids only if needed Mobilization Pain management by epidural cannula Discussion of the ERAS protocol Pancreatin capsules per os before eating
  Postoperative day 2:
  - Mobilization: As much as possible, autonomous movement
  Postoperative day 3:
  Ending epidural infusion cannula removal Mobilization as independently as possible
  Pain relief: oxycodone/naloxone p.o. to keep mobilization possible:
  Postoperative day 4:
  Support and encouragement continues Pain management at a level that allows mobility
  Arms: Enchanced recovery after surgery protocol

SUMMARY:
In the study, the enhanced recovery after surgery (ERAS) program is applied to total pancreatectomy (TP) and low-risk pancreaticoduodenectomy (PD) patients identified by a small number of acinar cells in the cut edge of the pancreas. The research setting is randomized and controlled. All patients arriving at the Tampere University Hospital (TAUH) for PD or TP surgery are recruited into the study. Recruited patients are randomized to the ERAS protocol and to the standard protocol recovery program. The ERAS program differs from the normal care protocol preoperatively, intraoperatively and postoperatively as explained in the following section.

In the ERAS protocol, both on the previous day of the surgery and on the following days, the patient is discussed with the patient about the benefits of the protocol used and the recovery program objectives. The purpose is to motivate and encourage the patient. On the day of surgery, the patient's intake of food and fluids is allowed to be closer to the surgery and the patient is also given a carbohydrate drink two hours before surgery. The nasogastric tube set at the beginning of surgery is removed at the end of the surgery and peripancreatic or perihepatic drains are not routinely placed. After surgery, drinking is allowed after four hours and the patient is encouraged to move as actively as possible in the bed. On the first and second postoperative day, the patient is allowed to enjoy normal food and drink according to his or her ability, and pancreatic capsules are given in the course of food. Additionally, the analgesic to be administered through the epidural cannula is dosed as far as possible to allow mobilization of the patient. The discussion on the benefits and recovery targets of the ERAS protocol are continued. On the third postoperative day, the epidural infusion is discontinued and the pain medication is moved to opioid-based pain management. This is continued until specific criteria for passing to the follow-up care are met.

Typical complications (pancreatic fistula, delayed gastric emptying, postpancreatectomy hemorrhage) are registered during hospitalization and their severity ratings according to ISGPS, ISPGF and Clavien-Dindo classifications are also determined. Other variables registered are the number of intensive care days, situations requiring new surgeries, 30 and 90 day mortality, the completion time of the criteria for passing to follow up care, and the total length of hospitalization. In addition, the need for readmissions is registered. The implementation of the ERAS protocol is followed by a separate tracking template, in which the nurses record the progress of the goals specified in the protocol on a daily basis. The results of the study are analyzed with the intention-to-treat principle.

DETAILED DESCRIPTION:
In the study, the enhanced recovery after surgery (ERAS) program is applied to total pancreatectomy (TP) and low-risk pancreaticoduodenectomy (PD) patients identified by a small number of acinar cells in the cut edge of the pancreas. The research setting is randomized and controlled. All patients arriving at the Tampere University Hospital (TAUH) for PD or TP surgery are recruited into the study. Patients will be sent a handout of the study along with the letter of invitation for the surgery itself. Recruitment takes place at the first appointment of the surgery where the surgeon presents the study to the patient. If the patient wishes to participate in the study, the patient issues a signature on the consent form. They are randomized to this ERAS program for shortened recovery period and a standard protocol recovery program. Allocation to the groups takes place using opaque envelope-coded randomization codes. The research nurse prepares the envelopes in twelve patient randomization blocs.

To determine the low risk PD-patients recruited, the pathologial sample of the cut-edge of the pancreas is analyzed by pathologist during the surgery. If the pancreatic cut-edge contains less than 40% acinar cells, the patients is considered low risk patient. This method is based on earlier studies in our pancreatic research group. All TP patients are per se in the small complication risk group. Only those patients with a low risk of complications continue to be involved in the study in standardized or ERAS protocol groups according to the original allocation.

ERAS protocol consist of following actions in comparison to standard protocol:

First appointment:

- Enlightenment on the benefits and objectives of the ERAS protocol

Call to the patient day before the surgery:

* Discussing the course, benefits and goals of care in ERAS
* 4 dl PreOp drink before bedtime

Operation day:

* Fluid intake allowed 2 hours before surgery
* 2 dl PreOP drink 2 h before cutting

Intraoperative:

* Drains in the peripancreatic or perihepatic regions are not set unless the surgeon sees this particular reason
* The nasogastric tube is removed at the end of the surgery

Postoperative:

* Mobilization with nurses assisted, possibly sitting on the edge of the bed if possible
* Drinks allowed after 4h surgery

Postoperative day 1:

* Drinking and normal food by mouth according to the patient's capabilities
* Removal of urinary catheter
* Intravenous liquids only if needed
* Mobilization physiotherapist and nurse guided as actively as possible
* Pain management by epidural cannula at the level to make mobilization possible
* Discussion of the ERAS protocol (objectives, benefits, time of passing to follow up care) (also continues on the following days) and encouragement
* If drains are set: amylase tests
* Pancreatin capsules per os before eating, 25,000 IU 1-2 capsules on big meals and 1 on snack (continued on the following days)

Postoperative day 2:

- Mobilization: As much as possible, autonomous movement

Postoperative day 3:

* Ending epidural infusion, cannula removal later if p.o. medication is sufficient
* As independent as possible

Pain relief: oxycodone / naloxone p.o. to keep mobilization possible:

1. 2x 5 / 2.5 mg ≤ 60 kg
2. 2x 10/5 mg> 60 kg
3. 2x 15 / 7.5> 100kg. In addition, paracetamol 1g three times a day p.o.

Postoperative day 4:

* Support and encouragement continues
* Pain management at a level that allows mobility
* Passing to follow up care when following criteria are met:

  1. The patient should be able to enjoy at least two meals without significant nausea
  2. Bowel movements returned
  3. The patient should be able to move, urinate, and perform daily operations at pre-operative level
  4. The patient does not need strong analgesics when moving
  5. The temperature, pulse rate, blood pressure and respiratory rate should be in the reference range or pre-cut level.
  6. The patient has no signs of bleeding.
* Pain medication changes to tramadol 100 mg three times a day when discharged

For all those involved in the study, PD's surgery technique is standardized to classic Whipple surgery, submersion bowel-pancreatic seam, antecholic gastro-jejunostomy and entero-entero anastomosis.

The patient is left out of the study if a patient is undergoing another surgery than PD, TP or does not undergo surgery at all. Likewise, the study is suspended from the consideration of the surgeon if, for any other reason, the patient may be expected to be a high complication risk patient.

Typical complications (pancreatic fistula, delayed gastric emptying, postpancreatectomy hemorrhage) are registered during hospitalization and their severity ratings according to ISGPS, ISPGF and Clavien-Dindo classifications are also determined. Other variables registered are the number of intensive care days, situations requiring new surgeries, 30 and 90 day mortality, the completion time of the criteria for passing to follow up care, and the total length of hospitalization. In addition, the need for readmissions is registered. The implementation of the ERAS protocol is followed by a separate tracking template, in which the nurses record the progress of the goals specified in the protocol on a daily basis. The results of the study are analyzed with the intention-to-treat principle.

The main variable of the study is the treatment period at the university hospital. The side variables are the total treatment time, the total amount of complications, and the number of readmissions. The hypothesis is that recovery is faster in the ERAS group, but the occurrence of complications and readmissions are the same in both groups.

A statistical power calculation, assuming 80% statistical power (1-β) and 5% significance level (α), was carried out with a continuous outcome superiority trial. The sample size was calculated using the main coefficient of variation assuming that in the standard protocolled patients the median of the discharge time is nine days and in the ERAS program for seven days, i.e. a presumption of approximately 20% decrease in treatment days. Three days were assumed to be the standard deviation. The sample size thus obtained is 36 per group, which is rounded up to approximately 80 patients in total.

When evaluating the time spent collecting the data, it is assumed that 20% of the patients will drop out of the study for various reasons. In TAUH, approximately 100 PDs and 15 TP patients are operated in two years and approximately 70% of patients of PD are in a low risk of complications. Consequently, the number of patients to be collected in two years would be approximately 0.7 ∙ 0.8 ∙ 100 + 0.8 ∙ 15 ≈ 68, which is almost sufficient for the purpose of this study to achieve statistical significance. The estimated duration of the study is therefore little more than two years. However, the study will be continued as long as necessary to collect the required number of patients. When half of the final number of patients has been collected, an interim analysis is made of the differences in the groups. If the results of the ERAS protocol are at least as good as the standard group, the study will be continued.

All recruited patients are asked for written consent for participation in the study. The research file is stored in the TAUH research register. Patient information and research results are treated confidentially in the manner required by the Finnish Personal Data Act. The final research results are reported at group level and the identification of individual investigators is not possible. The research funding is provided by the Tampereen Pancreatic Research Group the largest funders being the State Research Fund and Sigrid Jusélius Foundation. Also Finnish Medicine Foundation in providing personal funding.

The research has been approved by the Ethics Committee of the Tampere University Hospital. The earlier ERAS studies have shown that their use is safe and in most cases beneficial to the patient. In this study, it is novel that only small complication risk patients are included in the study. In addition, halfway between the research is performed an interim analysis to ensure the safety of the ERAS protocol. Patient's own consent is asked before surgery, and information on the research is provided within the limits of the success of the study. Patient's refusal or suspension of study does not affect the patient's treatment in any way.

ELIGIBILITY:
Inclusion Criteria:

* All PD or TP patients 18-99 years old

Exclusion Criteria:

* Any other surgery than PD or TP
* High risk patients
* Refusal for the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Days until discharge from university hospital | Up to 24 weeks
  Time in days since the entry to hospital on the surgery day to the discharge day to follow up care or home

SECONDARY OUTCOMES:
Days until discharge from follow up care | Up to 24 weeks
  Time in days since the entry to hospital on the surgery day to the discharge day from the follow up care
Total number of complications | Postoperatively up to 24 weeks
  Total number of postoperative complications
Readmission frequency | From the discharge up to 24 weeks for any cause related to surgery
  Number of readmissions in contrast to total patient number

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Laukkarinen, MD-PhD, Study Director — Dept. of Gastroenterology and Alimentary Tract Surgery, Tampere University Hospital, Finland
Locations (1):
- Tampere University Hospital Deparment of Gastroenterologic Surgery, Tampere, Finland